CLINICAL TRIAL: NCT02994355
Title: HIV Testing at Family Planning Clinics in Mombasa County, Kenya: A Cluster-Randomized Trial Comparing the Systems Analysis and Improvement Approach (SAIA) to Usual Procedures
Brief Title: HIV Testing at Family Planning Clinics in Mombasa County, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Nairobi (Other); Kenyatta National Hospital (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Ministry of Health, Mombasa County (Other Government)
Responsible Party: Principal Investigator, Scott McClelland, Professor, Medicine, Epidemiology, and Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00001851; 1K24HD088229-01 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: Family planning clinics; Implementation Science; Systems Analysis and Improvement Approach (SAIA)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Clinics (Experimental): Clinics randomized to the intervention will be introduced to the Systems Analysis and Improvement Approach (SAIA) to understand barriers to HIV testing in family planning clinics. Sequential process flow mapping will be used to highlight areas for improvement and then specific interventions will be implemented for the clinics with the goal of increasing HIV testing rates.
  Interventions: Other: Systems Analysis and Improvement Approach
- Control Clinics (No Intervention): Clinics randomized to the control arm of the study will continue HIV testing as per usual procedures.

INTERVENTIONS:
Other: Systems Analysis and Improvement Approach — 1. Understanding the cascade from FP clinic enrollment to HIV testing
  2. Use process mapping to identify modifiable bottlenecks
  3. Define and implement workflow adaptations to eliminate modifiable bottlenecks
  4. Monitor change in performance
  5. Repeat the analysis and improvement cycle (steps 1-4)
  Other Names: SAIA
  Arms: Intervention Clinics

SUMMARY:
Location: Family Planning Clinics in Mombasa County, Kenya

Introduction:

Integration of HIV treatment and prevention with family planning (FP) services is a promising approach for optimizing delivery of comprehensive healthcare for HIV-positive women, as well as prevention services for those who are negative. In Mombasa County, the USAID-supported AIDS Population and Health Integrated Assistance II Program revised the FP Clinic Register to capture HIV testing in 2008. However, the rate of HIV testing in FP clinics remains low. Our overarching objective is to assess the effectiveness, costs, and budget impact of implementing the systems analysis and improvement approach (SAIA) to increase HIV testing in FP clinics in Mombasa County.

Methods:

The investigators aim to conduct a cluster-randomized trial comparing the effect of the SAIA approach versus usual procedures on rates of HIV testing in first-time attendees at 20 intervention versus 20 control FP clinics in Mombasa County. The investigators will compare HIV testing rates for first-time FP clinic attendees in SAIA intervention versus control facilities after an additional year, during which FP clinics in the intervention arm will be encouraged to continue to use the SAIA tools with minimal support from the study team as the Mombasa County Ministry of Health will take ownership of implementation. Lastly, the investigators aim to estimate the incremental cost and budget impact of applying SAIA versus standard of care using an activity-based approach.

Anticipated Results:

The investigators anticipate that SAIA will produce significant and sustained improvement in HIV-testing rates in first-time FP clinic attendees in intervention clinics compared to control facilities. The use of a rigorous study design will provide strong evidence to guide integration of HIV testing into FP services in a wide range of settings. The inclusion of costing and budget impact analyses will assist policy makers in reaching informed decisions about implementation.

Anticipated Conclusion:

By addressing the crucial first step in the linkage of HIV and FP services, this research holds considerable promise for improving women's health by opening the gateway to HIV care and prevention.

DETAILED DESCRIPTION:
Integration of HIV treatment and prevention with family planning (FP) services is a promising approach for optimizing delivery of comprehensive healthcare for HIV-positive women, as well as prevention services for those who are negative. The need for integration of services is evident in Africa, which bears a disproportionate burden of HIV, high birth rates, and maternal mortality. A high and increasing proportion of African women use FP services, making this a potentially efficient venue for reaching them.

Testing for HIV is the gateway to care and prevention. Integrating HIV testing into FP clinics could open this essential gateway, decreasing stigma associated with seeking HIV testing while reducing costs. The antenatal setting provides a useful example. In many African countries, testing for HIV in antenatal clinics (ANCs) has become routine. Diagnosis of HIV during pregnancy has paved the way to substantial reductions in mother-to-child transmission of HIV and AIDS-related deaths in women of reproductive age. These achievements demonstrate the feasibility and impact of wide-scale HIV testing through existing reproductive health services. In contrast to ANCs, integration of HIV testing into FP services remains at a formative stage in much of Africa. Recent reviews support the feasibility of integrating these services, but invariably conclude that additional research is needed.

In Kenya, the National AIDS and STD Control Program (NASCOP) states that the FP clinic is a setting in which, "Failure to offer HIV testing and counseling is unacceptable, and will be considered negligent." However, there has been almost no operational assessment of HIV testing in Kenyan FP clinics. In Mombasa County, the USAID-supported AIDS Population and Health Integrated Assistance II Program revised the FP Clinic Register to capture HIV testing in 2008. However, the rate of HIV testing in FP clinics remains low, and the County has requested our assistance in addressing this prevention gap. Colleagues at the University of Washington Department of Global Health have developed a systems analysis and performance enhancement approach, using industrial and systems engineering techniques, that the investigators believe will be useful in this setting. The overarching objective is to assess the effectiveness, costs, and budget impact of implementing this systems analysis and improvement approach (SAIA) to increase HIV testing in FP clinics in Mombasa County. The investigators specific aims are as follows:

AIM 1: To conduct a cluster-randomized trial comparing the effect of the SAIA approach versus usual procedures on rates of HIV testing in first-time attendees at 12 intervention versus 12 control FP clinics in Mombasa County, Kenya.

HYP 1: After one year of study team support implementing SAIA vs. usual procedures, a higher proportion of first-time FP clinic attendees will be tested for HIV at intervention compared to control facilities

AIM 2: To determine whether the SAIA training results in a lasting effect, the investigators will compare HIV testing rates for first-time FP clinic attendees in SAIA intervention versus control facilities after an additional year, during which FP clinics in the intervention arm will be encouraged to continue to use the SAIA tools with minimal support from the study team. The Mombasa County Ministry of Health will take ownership of implementation during this phase.

HYP 2: After an additional year with minimal support from the study team, there will continue to be significantly higher rates of HIV testing in first-time FP clinic attendees at intervention compared to control facilities.

AIM 3: To estimate the incremental cost and budget impact of applying SAIA versus standard of care. Using an activity-based approach, the investigators will perform a costing analysis, estimating cost per new HIV diagnosis, both during active support from the study team and after a period without active support. The investigators will also estimate cost to scale up, and conduct a budget impact analysis from a Department of Health (DOH) perspective.

Expected Outcome and Significance:

The investigators anticipate that the SAIA approach will produce significant and sustained improvement in HIV-testing rates in first-time FP clinic attendees in intervention clinics compared to control facilities. The use of a rigorous study design to evaluate this scalable approach will provide strong evidence to guide integration of HIV testing into FP services in a wide range of settings. The inclusion of costing and budget impact analyses will assist policy makers in reaching informed decisions about implementation. By addressing the crucial first step in the linkage of HIV and FP services, this research holds considerable promise for improving women's health by opening the gateway to HIV care and prevention. Preliminary data on linkage to care and prevention services will inform development of future grant proposals.

ELIGIBILITY:
Inclusion Criteria for in-depth interviews:

* Adult family planning clinic staff
* If staff younger than 18 are encountered, they will be allowed to participate only if they qualify as emancipated minors in Kenya (14 years or older and married or pregnant).
* Able to provide written informed consent for in-depth interviews

Inclusion criteria for FP clinics in Mombasa:

-Clinics providing assent for participation in both the preliminary review and randomizations

Exclusion Criteria for FP clinics:

* Clinics planning to be closed during the study period
* Clinics unwilling to be randomized or to participate in the SAIA intervention/approach

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond S McClelland, MD, MPH, Principal Investigator — Professor of Medicine, Epidemiology, Global Health
Locations (24):
- Kenya (24):
  - Alfarooq, Mombasa
  - Jocham, Mombasa
  - Junda Dispensary, Mombasa
  - Junda, Mombasa
  - Kongowea, Mombasa
  - Magongo, Mombasa
  - Marimani, Mombasa
  - Mbuta, Mombasa
  - Mikindani, Mombasa
  - Mlaleo, Mombasa
  - Mrima, Mombasa
  - Mvita, Mombasa
  - Mwakirunge, Mombasa
  - Mwangaza, Mombasa
  - Pandya, Mombasa
  - Roadside, Mombasa
  - ShikaAdabu, Mombasa
  - Shukurani, Mombasa
  - Singawa, Mombasa
  - St. Thomas, Mombasa
  - Tudor, Mombasa
  - Waweni, Mombasa
  - Wema, Mombasa
  - Ziwa la ngombe, Mombasa

REFERENCES:
- [Background] WHO, UNFPA, IPPF, UNAIDS, UCSF. Sexual and reproductive health and HIV linkages: evidence review and recommendations. Geneva: 2009.
- [Background] UNAIDS. Global Report: UNAIDS Report on the Global AIDS Epidemic 2013. Geneva: 2013.
- [Background] National Department of Health South Africa, Medical Research Council South Africa, Human Sciences Research Council South Africa. South African demographic and health survey (SADHS). 2003.
- [Background] Uganda Bureau of Statistics, MEASURE DHS. Uganda demographic and health survey. 2011.
- [Background] Central Statistical Office Zambia, Ministry of Health Zambia, Tropical Diseases Research Centre Zambia, University Teaching Hospital Virology Laboratory Zambia, University of Zambia, The DHS Program II. Zambia Demographic and Health Survey 2013-14: Preliminary Report. Rockville, MD: 2014 September 2014.
- [Background] Oberzaucher N, Baggaley R. HIV voluntary counselling and testing: a gateway to prevention and care. Geneva, Switzerland: UNAIDS, 2002 June, 2002.
- [Background] Kenya National Bureau of Statistics, Ministry of Health Kenya, National AIDS Control Council, Kenya Medical Research Institute, National Council for Population and Development Kenya. Kenya Demographic and Health Survey 2014: Key Indicators. Nairobi, Kenya: 2015 March 2015.
- [Background] National AIDS/STD Control Programme MoPHaS. Guidelines for HIV testing and counselling in Kenya. Nairobi: NASCOP, 2008.
- [Background] Bloom DE. 7 billion and counting. Science. 2011 Jul 29;333(6042):562-9. doi: 10.1126/science.1209290. PMID 21798935
- [Background] Hogan MC, Foreman KJ, Naghavi M, Ahn SY, Wang M, Makela SM, Lopez AD, Lozano R, Murray CJ. Maternal mortality for 181 countries, 1980-2008: a systematic analysis of progress towards Millennium Development Goal 5. Lancet. 2010 May 8;375(9726):1609-23. doi: 10.1016/S0140-6736(10)60518-1. Epub 2010 Apr 9. PMID 20382417
- [Background] Lozano R, Wang H, Foreman KJ, Rajaratnam JK, Naghavi M, Marcus JR, Dwyer-Lindgren L, Lofgren KT, Phillips D, Atkinson C, Lopez AD, Murray CJ. Progress towards Millennium Development Goals 4 and 5 on maternal and child mortality: an updated systematic analysis. Lancet. 2011 Sep 24;378(9797):1139-65. doi: 10.1016/S0140-6736(11)61337-8. Epub 2011 Sep 19. PMID 21937100
- [Background] Lindegren ML, Kennedy CE, Bain-Brickley D, Azman H, Creanga AA, Butler LM, Spaulding AB, Horvath T, Kennedy GE. Integration of HIV/AIDS services with maternal, neonatal and child health, nutrition, and family planning services. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD010119. doi: 10.1002/14651858.CD010119. PMID 22972150
- [Background] Kennedy CE, Spaulding AB, Brickley DB, Almers L, Mirjahangir J, Packel L, Kennedy GE, Mbizvo M, Collins L, Osborne K. Linking sexual and reproductive health and HIV interventions: a systematic review. J Int AIDS Soc. 2010 Jul 19;13:26. doi: 10.1186/1758-2652-13-26. PMID 20642843
- [Background] Spaulding AB, Brickley DB, Kennedy C, Almers L, Packel L, Mirjahangir J, Kennedy G, Collins L, Osborne K, Mbizvo M. Linking family planning with HIV/AIDS interventions: a systematic review of the evidence. AIDS. 2009 Nov;23 Suppl 1:S79-88. doi: 10.1097/01.aids.0000363780.42956.ff. PMID 20081392
- [Background] Madon T, Hofman KJ, Kupfer L, Glass RI. Public health. Implementation science. Science. 2007 Dec 14;318(5857):1728-9. doi: 10.1126/science.1150009. No abstract available. PMID 18079386
- [Background] Glasgow RE, Vinson C, Chambers D, Khoury MJ, Kaplan RM, Hunter C. National Institutes of Health approaches to dissemination and implementation science: current and future directions. Am J Public Health. 2012 Jul;102(7):1274-81. doi: 10.2105/AJPH.2012.300755. Epub 2012 May 17. PMID 22594758
- [Background] UNAIDS. The GAP Report. Geneva: Joint United National Programme on HIV/AIDS (UNAIDS), 2014.
- [Derived] Thomas D, Wanje G, Eastment MC, McClelland RS, Mwaringa E, Patta S, Jaoko W, Kinuthia J, Abubakar A, Sherr K, Barnabas RV. The cost of implementing the Systems Analysis and Improvement Approach for a cluster randomized trial integrating HIV testing into family planning services in Mombasa County, Kenya. BMC Health Serv Res. 2022 Dec 5;22(1):1480. doi: 10.1186/s12913-022-08828-z. PMID 36471311
- [Derived] Long JE, Eastment MC, Wanje G, Richardson BA, Mwaringa E, Mohamed MA, Sherr K, Barnabas RV, Mandaliya K, Jaoko W, McClelland RS. Assessing the sustainability of the Systems Analysis and Improvement Approach to increase HIV testing in family planning clinics in Mombasa, Kenya: results of a cluster randomized trial. Implement Sci. 2022 Oct 4;17(1):70. doi: 10.1186/s13012-022-01242-3. PMID 36195890
- [Derived] Eastment MC, Long JE, Wanje G, Richardson BA, Mwaringa E, Sherr K, Barnabas RV, Mandaliya K, Jaoko W, McClelland RS. Qualitative evaluation of the Systems Analysis and Improvement Approach as a strategy to increase HIV testing in family planning clinics using the Consolidated Framework for Implementation Research and the Implementation Outcomes Framework. Implement Sci Commun. 2022 Sep 8;3(1):97. doi: 10.1186/s43058-022-00342-x. PMID 36076250

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Family Planning Clinics
Period: Overall Study
Arm/Group | Intervention Clinics | Control Clinics
Started | NA; 12 Family Planning Clinics (Data was collected at the clinic level. Data was collected at the clinic level.) | NA; 12 Family Planning Clinics (Data was collected at the clinic level. Data was collected at the clinic level.)
Completed | NA; 11 Family Planning Clinics (Data was collected at the clinic level. Data was collected at the clinic level.) | NA; 11 Family Planning Clinics (Data was collected at the clinic level. Data was collected at the clinic level.)
Not Completed | NA; 1 Family Planning Clinics | NA; 1 Family Planning Clinics

BASELINE CHARACTERISTICS:
Population: These are descriptions of entire family planning clinics.
Units Other Than Participants: Family Planning Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Clinics | Control Clinics | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Family Planning Clinics) | 12 | 11 | 23
Age, Categorical [Count of Units; unit: Family Planning Clinics]
  <=18 years | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: Family Planning Clinics]
  Female | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Units; unit: Family Planning Clinics]
  American Indian or Alaska Native | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Data was collected at the clinic level. | NA — Data was collected at the clinic level. | NA — Total not calculated because data are not available (NA) in one or more arms.
Public Clinic [Count of Units; unit: Family Planning Clinics] | 6 | 6 | 12
Urban Clinic [Count of Units; unit: Family Planning Clinics] | 4 | 4 | 8
Complete auditory privacy [Count of Units; unit: Family Planning Clinics] | 7 | 7 | 14
Complete visual privacy [Count of Units; unit: Family Planning Clinics] | 8 | 6 | 14
FP clinic manager aware of most recent National HIV Guidelines [Count of Units; unit: Family Planning Clinics] | 6 | 9 | 15
Number of FP providers trained in HTC [Median (Inter-Quartile Range); unit: Family Planning Clinics] | 1 [0 to 2] | 1 [0 to 2] | 1 [0 to 2]
Clients required to pay for HIV testing [Count of Units; unit: Family Planning Clinics] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible (Not Known HIV+) New FP Clients Who Are Tested for HIV in the Months 9-12 of the Study in Intervention and Control Facilities
Time Frame: Months 9-12 of the study
Population: Data was collected at the clinic level.
Measure: Mean (Standard Deviation); unit: Percentage tested for HIV
Units Other Than Participants: FP Clinics
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | NA | NA
Number analyzed (FP Clinics) | 12 | 11
Percentage tested for HIV | 42 (26) | 32 (15)
Statistical Analysis 1: Comparison: Intervention Clinics vs Control Clinics; Test type: Superiority; p < 0.05, Poisson Regression; Prevalence rate ratio = 1.33, 95% CI 2-sided [1.16 to 1.52]

2. Secondary Outcome: Percentage of New FP Clients Who Are Counseled About HIV Testing in the Months 9-12 of the Study in Intervention and Control Facilities, Adjusted for Baseline
Time Frame: Months 9-12 of the study
Population: Data was collected at the clinic level.
Measure: Mean (Standard Deviation); unit: Percentage counseled for HIV
Units Other Than Participants: FP Clinics
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | NA | NA
Number analyzed (FP Clinics) | 12 | 11
Percentage counseled for HIV | 85 (27) | 67 (34)
Statistical Analysis 1: Comparison: Intervention Clinics vs Control Clinics; Test type: Superiority; p < 0.05, Poisson regression; Prevalence rate ratio = 1.27, 95% CI 2-sided [1.15 to 1.30]

3. Secondary Outcome: Percentage of New FP Clients Who Are Tested for HIV After Year of Minimal Support
Time Frame: Months 13-24 of the study
Population: Data was collected at the clinic level.
Measure: Mean (Standard Error); unit: % tested for HIV
Units Other Than Participants: FP Clinics
Arm/Group | Intervention Clinics | Control Clinics
Number analyzed (Participants) | NA | NA
Number analyzed (FP Clinics) | 12 | 11
% tested for HIV | 61 (7) | 19 (6)
Statistical Analysis 1: Comparison: Intervention Clinics vs Control Clinics; Test type: Superiority; p < 0.05, Poisson regression; Prevalence rate ratio = 3.23, 95% CI 2-sided [2.29 to 4.55]

ADVERSE EVENTS:
Time Frame: 2 years
Description: All cause mortality was not assessed.
Arm/Group | Intervention Clinics | Control Clinics
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
First, increases in HTC could not be independently verified through direct observation of HIV counseling sessions or through increases in consumption of HIV testing commodities. Second, due to collinearity, it was not possible to adjust for baseline differences in HIV testing as planned for this analysis. Lastly, this intervention focused on HIV testing, and did not extend to additional steps in the HIV prevention and care cascades.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT02994355/Prot_SAP_000.pdf